CLINICAL TRIAL: NCT05914363
Title: Evaluating the Impact of an Improved Household Flooring Intervention on Enteric and Parasitic Infections in Rural Settings in the Counties of Bungoma and Kwale, Kenya
Brief Title: Evaluating Impact of Improved Floors on Health
Acronym: SABABU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Jomo Kenyatta University of Agriculture and Technology (Other); International Centre of Insect Physiology and Ecology (ICIPE) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 28307; 424/4 (Other: KEMRI SERU)
Record Dates: First submitted 2023-04-05; First posted 2023-06-22 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-06

CONDITIONS: Diarrhoeal Disease; Hookworm Infection; Ascaris Lumbricoides Infection; Trichuris Infection; Tungiasis
MeSH Terms: conditions — Hookworm Infections; Trichuriasis; Tungiasis | interventions — Albendazole; Therapeutics

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (improved floor) (Experimental): * Replacement of rudimentary floors with an improved floor,
  * Support for behaviour change through 'floor clubs'.
  * Annual mass treatment for STH infections (400 mg albendazole)
  * Treatment of tungiasis in those affected by heavy infections (at 0 and 12 months) according to county DoH recommendations
  Interventions: Other: Sealed washable floor plus behaviour change; Behavioral: Behaviour change intervention; Drug: Routine deworming; Procedure: treatment for tungiasis
- Control (rudimental floor) (Active Comparator): * Annual mass treatment for STH infections (400 mg albendazole)
  * Treatment of tungiasis in those affected by heavy infections (at 0 and 12 months) according to county DoH recommendations
  Interventions: Drug: Routine deworming; Procedure: treatment for tungiasis

INTERVENTIONS:
Other: Sealed washable floor plus behaviour change — Replacement of rudimentary floors with a cement stabilised floor in all rooms in the dwelling
  Arms: Intervention (improved floor)
Behavioral: Behaviour change intervention — Support for behaviour change through 'floor clubs' and the provision of printed guides
  Arms: Intervention (improved floor)
Drug: Routine deworming — Treatment of all household members for STH infections (400 mg albendazole in those aged 24 months and above; 200 mg albendazole in those aged 12-23 months)
  Other Names: albendazole
Procedure: treatment for tungiasis — Treatment of tungiasis in those affected by heavy infections (at 0 and 12 months) according to county Department of Health recommendations

SUMMARY:
The goal of this intervention study is to learn about the impact of household flooring on health in rural Kenya, and test whether providing an improved (cement stabilised, washable) floor improves the health of children and their care providers.

The main questions the study aims to answer are:

* What is the effect of providing a sealed, washable floor on the prevalence of infections that cause diarrhoea, intestinal worms and sand flea infections?
* To what extent does the intervention reduce contamination of floors with pathogens within the home?
* What is its effect of the intervention on the wellbeing of caregivers and children?
* Over the course of a year, do the new floors remain undamaged, with no cracks?
* Do participants living with the new floors, and the masons that helped to install the floors, like them and feel they are practical and affordable?

The study will involve a trial, where half of the recruited households will be randomly chosen to receive the new floor in addition to some support on how to care for the floor and keep it clean. The other half of households will not receive anything at first, but at the end of the research project will also receive a new floor.

Before the new floors are installed, the investigators will make several assessments in all study households. These will include a survey to measure household characteristics; a stool survey, to measure how many people are infected with diarrhoea-causing microorganisms and parasitic worms; a jigger flea examination among children; wellbeing assessments among children and caregivers; and soil sampling to identify microorganisms on the floor of the household.

When households receive the new floor, participants will have to move out of their house for up to 7 days during installation. Participants will also be asked to attend some group meetings to discuss ways of taking care of the floor and keeping it clean.

Assessments will be repeated 12 months after the floor has been delivered, and additional interviews will be held with a small number of randomly selected participants. Throughout the 12 months following delivery of the intervention, investigators will make unannounced visits to households to check the condition of the floor. Participants will also be offered treatment for parasitic worm infections after assessments have been completed at the start and end of the project.

DETAILED DESCRIPTION:
Earthen floors are often damp or dusty and difficult to clean, providing an ideal environment for faecal pathogens and parasites. Cross-sectional studies have revealed associations between household flooring and health outcomes, but robust experimental evidence is scant. This study will evaluate the impact of an improved household flooring intervention on enteric infections, soil-transmitted helminth (STH) infections, and tungiasis through implementation of a cluster-randomised trial in two rural settings in Kwale and Bungoma Counties, Kenya.

The primary aim of this study is to evaluate the effectiveness of an improved flooring intervention in reducing the burden of enteric infections, STH and tungiasis in participating households through implementation of a randomised controlled trial (RCT) in two distinct settings in rural Kenya. The primary objectives are to quantify impact on the prevalence of enteric infections, STH infections, and tungiasis. Secondary objectives include assessing impact on the wellbeing of caregivers and children, self-report gastrointestinal illness in children, and the extent to which entero-pathogen and parasitic contamination of floors is reduced within the home. We will also examine the differential effects across community and household contexts (including water, sanitation, and hygiene (WASH) infrastructure, animal husbandry, user adherence and study site). Lastly, we deliver a process evaluation to determine the practicality, acceptability, costs, and durability of the improved flooring intervention and how environmental, installation, and use factors affect these.

In total, 440 clusters (households) across both sites are allocated to either control or intervention group, in which a low-cost, sealed, washable cement-based floor is installed in all eligible buildings of the dwelling, alongside a floor care guide provided during an induction meeting. Prevalence of enteric infections in children under 5 years will be assessed via stool surveys and PCR; prevalence of tungiasis infection in children 1-14 years based on clinical exam; and prevalence of STH infection in all household members over 1 year assessed via Kato-Katz. Following the 12-month implementation period and final assessments, control households will be offered improved floors.

ELIGIBILITY:
Inclusion Criteria:

* Household with a child under 5 years of age that meets structural criteria (unimproved earthen flooring throughout, structurally sound), with members willing to temporarily relocate.

Exclusion Criteria:

* Households that are intending to move within the next 12 months, or that have improved flooring in any rooms or are not structurally sound.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2200 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Enteric infections | 12 months
  Prevalence of enteric infections (detected through PCR) in children under 5 years old will be assessed using cross-sectional stool surveys including all enrolled children under 5 years before installation of floors and 12 months after receiving the floors. Pathogens to be identified from those observed at baseline using a multipathogen panel on a subset of 100 samples.
Tungiasis infections | 12 months
  Prevalence of tungiasis (detected through clinical examination of hands and feet) in children under 15 years old will be assessed using cross-sectional clinical assessment surveys including all enrolled children under 15 years before installation of floors and 12 months after receiving the floors.
STH infections | 12 months
  Prevalence of at least one STH infection (hookworm, ascaris and trichuris infections; detected through kato katz) in all household members 12 months and older will be assessed using cross-sectional stool surveys including all enrolled people over 12 months of age before installation of floors and 12 months after receiving the floors.

SECONDARY OUTCOMES:
Gastrointestinal illness | 12 months
  Prevalence of gastrointestinal illness in children under 5 years - assessed in both study arms based on caregiver reported symptoms
Intensity and severity of tungiasis | 12 months
  Intensity of tungiasis and severity of acute and chronic tungiasis-associated pathology in children <15 years - assessed using clinical severity scores (range: 0-110, high scores indicating increased severity/worse outcome)
Quality of Life for children aged 8 to 14 years | 12 months
  Quality of Life assessed in children ages 8 to 14 years in both arms using the standardised EQ5D-Y (EuroQol 5-dimension health-related quality of life tool for children; values are anchored at 1 (full health) and 0 (a state as bad as being dead))
Quality of Life and subjective wellbeing in primary caregivers | 12 months
  Quality of Life assessed in primary caregivers in both arms using the standardised EQ5D tool (EuroQol 5-dimension health-related quality of life tool for adults; values are anchored at 1 (full health) and 0 (a state as bad as being dead))
Prevalence of Ascaris lumbricoides infection | 12 months
  Ascaris lumbricoides (roundworm) infection prevalence in all household members >1 year assessed using Kato Katz
Prevalence of hookworm infection | 12 months
  Hookworm infection prevalence in all household members >1 year assessed using Kato Katz
Prevalence of Trichuris trichiura infection | 12 months
  T. trichiura (whipworm) infection prevalence in all household members >1 year assessed using Kato Katz
Environmental contamination - enteric pathogens | 12 months
  Environmental contamination for human-specific and animal faecal markers - assessed from dust/soil samples from household cooking areas and living rooms using PCR.
Environmental contamination - tungiasis | 6 months
  Contamination of floors with eggs, larvae, pupae and adults of T. penetrans - assessed through entomology soil surveys

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pullan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Ulrike Fillinger, PhD, Principal Investigator — icipe; Charles Mwandawiro, PhD, Principal Investigator — Kenya Medical Research Institute; James Wambua KALULI, PhD, Principal Investigator — JKUAT
Locations (1):
- Dzombo ward, Kwale, Kwale County, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this study and underlying each article (text, tables, figures, and appendices), including quantitative, de-identified, individual participant data and a data dictionary, will be made available following publication of the article(s).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The quantitative, individual, de-identified, participant data that underlie the results reported in each published article (text, tables, figures, and appendices) will be made available within three months of publication of each article, with no end date.
Access Criteria: The data will be made available to members of the scientific and medical community for non-commercial use only, upon email request to the corresponding author. Written proposals will be assessed by members of the SABABU Trial Group and a decision made about the appropriateness of the use of data. Data will be stored at LSHTM Data Compass, the London School of Hygiene & Tropical Medicine digital data repository The data will be available to anyone who wishes to access the data through the LSHTM Data Compass, the London School of Hygiene & Tropical Medicine digital data repository.
  URL is https://datacompass.lshtm.ac.uk/

REFERENCES:
- [Derived] Halliday KE, Kepha S, Legge H, Allen E, Dreibelbis R, Elson L, Kakoi BK, Mcharo C, Muli S, Mwongeli J, Njomo D, Njoroge MM, Ochwal V, Oswald WE, Rono M, Safari TK, Filinger U, Kaluli JW, Mwandawiro CS, Pullan RL. Evaluating impacts of improved flooring on enteric and parasitic infections in rural households in Kenya: study protocol for a cluster-randomised controlled trial. BMJ Open. 2025 Jun 6;15(6):e090464. doi: 10.1136/bmjopen-2024-090464. PMID 40480665